CLINICAL TRIAL: NCT02816307
Title: Etiology of Endocarditis in Negative Blood Cultures
Acronym: ENDOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-39; 2012-A01549-34 (Other: ANSM)
Record Dates: First submitted 2016-06-21; First posted 2016-06-28 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Infective Endocarditis (IE)
MeSH Terms: conditions — Endocarditis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Infective endocarditis (Experimental)
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples

SUMMARY:
Infective endocarditis remains a serious disease that requires fast and specialized support in 2012. However, 24% of endocarditis unanswered etiology. The systematic use of new policy diagnosis, including (i) a systematic use of specific PCR techniques and (ii) the search for markers of inflammatory and tumoral diseases, should increase the number of positive etiological diagnosis of culture-negative samples.

Secondly, because of the seriousness of the disease, the investigators were led to develop a new score: score for admission. This score, realized in less than 4 hours from the admission of the suspected patient with endocarditis, should allow for immediate probabilistic antibiotic treatment after completion of the diagnostic kit. The modified Duke score give its results in 4 to 7 days. With the score of admission thus diagnostic processes are accelerated and, where appropriate, empirical antibiotic therapy started.

Primary: Evaluate the effectiveness of the new diagnostic strategy on etiological identification of endocarditis.

Secondary: Validate the "admission" score compared to the modified Duke score.

ELIGIBILITY:
Inclusion Criteria:

* Patient with endocarditis diagnostic kit prescribed
* Patient is more than 18 years old
* Patient who freely signed written informed consent.
* Patient affiliated to a health assurance

Exclusion Criteria:

* Minor patient (<18 years)
* Patient pregnant or breastfeeding
* Patient incapable or unable to consent
* Private patient of liberty or under court order
* Patient refusing to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3033 (Actual)
Dates: Start 2013-06-07 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with an etiological diagnosis of endocarditis | 6 years

SECONDARY OUTCOMES:
The "admission" score | 1 day
the Duke score | 1day

CONTACTS AND LOCATIONS:
Overall Officials: URIELLE DESALBRES, Study Director — Assistance Publique Hopitaux De Marseille; JEAN PAUL CASALTA, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assitance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No